CLINICAL TRIAL: NCT05419271
Title: Controlled Internal Convection in Low Flow Hemodialysis of Dialysate: Removal of Beta-2-microglobulin
Acronym: CIMHBaDD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-0017
Record Dates: First submitted 2022-05-16; First posted 2022-06-15 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-05

CONDITIONS: Daily Home Hemodialysis
Keywords: daily dialysis; home hemodialysis; Middle-molecular weight toxins; Beta2-microglobulin; Push-Pull

STUDY DESIGN:
Intervention Model Description: A prospective cross-over trial testing the efficiency of internal convection on Beta2-microglobulin in daily home hemodialysis, intradialytic fall of B2m levels is compared in 16 patients treated by one session of dialysis with 9L internal convection and one usual session with free internal convection.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental convection (Experimental): session of dialysis with 9L internal convection
  Interventions: Procedure: home hemodialysis session with 9L internal convection
- free internal convection (No Intervention): session of dialysis with free internal convection

INTERVENTIONS:
Procedure: home hemodialysis session with 9L internal convection — home hemodialysis session with 9L internal convection
  Arms: experimental convection

SUMMARY:
Since 2013 daily home hemodialysis allows low volumes of convection. This study is a prospective cross-over trial testing the efficiency of internal convection on Beta2-microglobulin in daily home hemodialysis.

DETAILED DESCRIPTION:
Daily home hemodialysis with low dialysate volume system does not normally allow convection. Middle molecular weight toxins clearance is therefore lower. Beta2-microglobulin is considered representative of these middle molecules and contributes to the uremic toxic state.

Since 2013 daily home hemodialysis allows low volumes of convection ranging from 0 to 9L per session. This technology is called "push pulls" and uses internal convection.

This study is a prospective cross-over trial testing the efficiency of internal convection on Beta2-microglobulin in daily home hemodialysis.

Intradialytic fall of B2m levels is compared in 16 patients treated by one session of dialysis with 9L internal convection and one usual session with free internal convection.

The Kt/V of urea, the phosphorus and sodium removal, the plasma fall of myoglobin, prolactin, kappa and lambda free light chains, intradialytic fall of orosomucoid will be compared between the two session as secondary objectives.

ELIGIBILITY:
Inclusion Criteria:

* home hemodialysis since at least 2 weeks
* hemodialysis since at least 3 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2022-05-09 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Middle molecular weight toxins clearance | during hemodialysis procedure
  Beta2-microglobulin levels

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Caen Normandie, Caen, France